CLINICAL TRIAL: NCT05904223
Title: Effect of IN Hospital PCR Based Assessment of Patients With Lower Respiratory Tract Infections on LEngth of Stay - INHALE Trial
Brief Title: Effect of IN Hospital PCR Based Assessment of Patients With Lower Respiratory Tract Infections on LEngth of Stay
Acronym: INHALE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexander Zoufaly (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor-Investigator, Alexander Zoufaly, PI, Klinik Favoriten
Organization: Klinik Favoriten (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: INHALE
Record Dates: First submitted 2023-05-23; First posted 2023-06-15 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Respiratory Infection
Keywords: Biofire
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): standard of care (SOC) group = control group:
  * Routine laboratory parameters (CBC, CRP, kidney and liver parameters, etc.) on the day of admission and when clinically necessary - decision is made by the physician in charge
  * Sputum microscopy for quality assessment (via Bartlett score)
  * Chest X-ray on the day of admission or the day after
  * 2 Sets of blood cultures (if temperature >38°)
  * Pneumococcus urine antigen test for every patient with proven or suspected pneumonia
  * Legionella urine antigen test for every patient with proven or suspected pneumonia and clinical suspicion for Legionella infection (travel history, air condition, elevated CK, hyponatremia, reduced kidney function)
  * Antibiotic treatment if deemed necessary by the treating physician
- Standard of Care + Respiratory Panel (Experimental): Pneumonia panel plus group = intervention group
  * Sputum analysis via the BIOFIRE® FILMARRAY® Pneumonia Panel plus
  * Routine laboratory parameters (CBC, CRP, kidney and liver parameters, etc.) on the day of admission and when clinically necessary - decision is made by the physician in charge
  * Sputum microscopy for quality assessment (via Bartlett score)
  * Chest X-ray on the day of admission or the day after
  * 2 Sets of blood cultures
  * Pneumococcus urine antigen test for every patient with proven or suspected pneumonia
  * Legionella urine antigen test for every patient with proven or suspected pneumonia and
  * Antibiotic treatment if deemed necessary by the treating physician
  Interventions: Diagnostic Test: Respiratory Panel PCR Sputum

INTERVENTIONS:
Diagnostic Test: Respiratory Panel PCR Sputum — Multiplex PCR Respiratory Panel from Biomerieux used on Patients Sputum
  Arms: Standard of Care + Respiratory Panel

SUMMARY:
Does the use of the BIOFIRE® FILMARRAY® Pneumonia Panel plus in hospitalized patients with lower respiratory infections lead to a reduction in length of hospital stay (LOS) and customized antibiotic treatment (higher amount of specific vs empiric treatment, shorter treatment duration, less antibiotic treatment, lower incidence of side effects) compared to the standard of care?

DETAILED DESCRIPTION:
Lower respiratory tract infections (LRTIs) like pneumonia, exacerbations of COPD or bronchitis are caused by several viral and/or bacterial pathogens. Even in huge epidemiological studies the causative pathogen can just be detected in approximately 50% of pneumonia cases. In clinical practice the pathogen is only known in few cases, e.g. Legionella via urine antigen test. It is impossible to distinguish the triggering bacteria by clinical parameters and even accurate differentiation between bacterial and viral infections is often not possible. The same problem exists for other LRTIs.

The lack of knowledge of the causative pathogen leads to several problems:

First, clinicians tend to observe patients after treatment initiation for a longer period than probably necessary, which may lead to an increased length of hospital stay. Secondly, the antibiotic treatment has to be broad enough to cover all possible pathogens empirically. This might lead to an overuse of broad-spectrum antibiotics, an increased risk of side effects, the development of antibiotic resistance or even delayed treatment of the causative agent. Finally, antibiotics are prescribed erroneously for viral infections, which have been misinterpreted as bacterial infections by clinicians.

The BIOFIRE® FILMARRAY® Pneumonia Panel plus can help to solve these problems by identifying the causative pathogen in LRTIs within 1.5 hours. The decision of the treatment and its duration would be pathogen driven and no longer just empirically based on a lot of unknown factors.

The investigators would like to perform the following study with two groups: standard of care (control group) vs Pneumonia panel plus (intervention group). Both groups will receive the standard of care treatment but the intervention group will additionally have their sputum analyzed via the BIOFIRE® FILMARRAY® Pneumonia Panel plus.

Additional information empiric vs specific treatment:

* empiric therapy - every antimicrobial therapy prescribed without knowing the pathogen

  o Amoxicillin/Clavulanic acid or Cefuroxime or Ceftriaxone/Cefotaxime or Piperacillin/Tazobactam or Levofloxacin
* Specific therapy - pathogen driven, prescribed knowing the pathogen; narrowed spectrum of agent

  * Pneumococcus - Penicillin G
  * H. influenzae - Cefuroxime or Doxycycline
  * Moraxella - Cefuroxime or Doxycycline
  * MSSA - Cefazolin or Flucloxacillin
  * MRSA - Linezolid or Vancomycin
  * Pseudomonas - Ceftazidime
  * E. coli - Cefuroxime or third generation Cephalosporin or Ciprofloxacin
  * Klebsiella - Cefuroxime or third generation Cephalosporin or Ciprofloxacin
  * Proteus, Serratia - third generation Cephalosporin or Ciprofloxacin
  * Enterobacter cloacae - Ertapenem
  * Legionella - Levofloxacin or Azithromycin
  * Mycoplasma - Azithromycin or Doxycycline
  * In case of ESBLs - Ertapenem or Meropenem
  * In case of carbapenemases - Ceftazidime/Avibactam (OXA48, KPC) or Meropenem/Vaborbactam (KPC) or Aztreonam +/- Ceftazidime/Avibactam (MBL +- others)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Hospitalised patients on a general ward
* Ability to give consent
* Ability to produce sputum

AND (one of the following diagnosis)

* acute exacerabation of COPD (defined as known COPD and worsening of symptoms like dyspnea +/- wheezing +/- increased sputum purulence and the need for additional treatment)
* Pneumonia (diagnosed via chest X-ray)

OR

Lower respiratory infection (which does not belong to one of the two former diagnosis) with following symptoms:

At least one criterion Cough (more than usual if smoker) Dyspnea Increased sputum purulence

AND (at least one criterion) Respiratory rate ≥22/min Reduced oxygen saturation (<95%) (or worsening of oxygen saturation by 3% (e.g. in patients with COPD) Fever (temp >38°C) Rales/wheezing Chest pain upon breathing

Exclusion Criteria:

* Other proven or suspected systemic diseases which require antibiotic treatment, like:

  * Intraabdominal infections (appendicitis, cholecystitis, diverticulitis, peritonitis)
  * C. difficile associated diarrhea (only if existing on admission otherwise it will be identified as a side effect)
  * Urinary tract infections like pyelonephritis, urosepsis, cystitis + fever (asymptomatic bacteriuria is NOT an exclusion criterion)
  * Acute bacterial skin and skin structure infections (erysipelas, abscess with systemic symptoms, diabetic foot infection, osteomyelitis)
  * Another single cause which can explain the respiratory symptoms better than an infection (acute heart failure, pulmonary embolism, hypertension induced lung edema)
* Proven respiratory infection via another PCR based system (e.g. influenza or tuberculosis)
* Inability to give consent
* Inability to produce sputum
* Moribund and palliative patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
length of stay (LOS) in days | From admission to discharge or death, whichever comes first, assessed up to 12 Months
  How long is the lenght of stay in days (half-days)?

SECONDARY OUTCOMES:
Duration of antibiotic treatment needed represented as days of treatment (DOT) | From start of antibiotic treatment to discontinuation of any cause, assessed up to 12 Months
  How long is the duration of antibiotic treatment in days?
Number of usage of specific vs empiric antibiotic treatment | From start of antibiotic treatment to discontinuation of any cause, assessed up to 12 Months
  Is there a difference in used antibiotic treatment?
Cost of antibiotic treatment | From start of antibiotic treatment to discontinuation of any cause, assessed up to 12 Months
  Is there a differnece in cost of antibiotic treatment?
In hospital and 30-day mortality | From admission to death or 30 days after admission
  Is there a difference in 30-day mortality?
C. difficile associated diarrhea within 30-day-follow-up | From admission to death or 30 days after admission
  Is there a diference in incidence of C. difficile associated diarrhea?
30-day re-admission rate | From admission to death or 30 days after admission
  Is there a difference in 30-day re-admission rate?

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zoufaly, Prof. Dr., Principal Investigator — Klinik Favoriten
Locations (1):
- Klinik Favoriten, Vienna, Österreich, Austria

IPD SHARING:
Plan to Share IPD: No